CLINICAL TRIAL: NCT03080896
Title: Comparison of Video-Laryngoscope Versus a Combination of a Video-Laryngoscope and Disposable Bronchoscope for Predicted Difficult Airway Intubation of Anesthetized Patients for Oral Cavity, Pharynx or Larynx Surgery
Brief Title: Video-Laryngoscope Alone or With Bronchoscope for Predicted Difficult Intubation
Acronym: COMBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Ambu A/S (Industry)
Responsible Party: Principal Investigator, Rainer Lenhardt, Professor, University of Louisville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #15.0096
Record Dates: First submitted 2017-01-27; First posted 2017-03-15 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Intubation; Difficult

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- control group videolaryngoscope/preformed stylet (Active Comparator): The control group will intubate using the video-laryngoscope / pre formed stylet. Will convert to using video-laryngoscope and fiber-optic bronchoscope (aScope III) if failure to intubate occurs
  Interventions: Device: King Vision video-laryngoscope with #3 disposable blade and endotracheal tube stylet; Device: fiberoptic bronchoscope aScope III
- Interventional Group videolaryngoscope/fibeoptic bronch (Experimental): The interventional group will Intubate using the video-laryngoscope and the fiber-optic bronchoscope (aScope III)
  Interventions: Device: fiberoptic bronchoscope aScope III

INTERVENTIONS:
Device: King Vision video-laryngoscope with #3 disposable blade and endotracheal tube stylet — intubation using King Vision video-laryngoscope with #3 disposable blade with stylet convert to intubation with video-laryngoscope and fiber-optic bronchoscope bronchoscope (aScope III) for failure to intubate after three attempts
  Other Names: Ambu aScope III
  Arms: control group videolaryngoscope/preformed stylet
Device: fiberoptic bronchoscope aScope III — Intubation using the videolaryngoscope/fiberoptic bronchoscope (aScope III)
  Other Names: aScope III by Ambu

SUMMARY:
Using a combination of the video-laryngoscope with the disposable fiber-optic bronchoscope (aScope III) is a feasible way to facilitate successful intubation in a timely manner, in patients with predicted difficult airway due to tumors in the oral cavity, pharynx or larynx To test the hypothesis that combination of video-laryngoscope with the fiber-optic bronchoscope is superior to video-laryngoscope alone for intubation of patients with oral cavity, pharyngeal or laryngeal pathologies undergoing surgery

DETAILED DESCRIPTION:
Detailed Description:

All subjects consented to this study will require endotracheal intubation. They will be randomly assigned to either one of two groups. The randomization will be stratified on whether the subject has an oral cavity/pharynx tumor or laryngeal tumor. The randomization groups are:

1. Intubation using King Vision video-laryngoscope with the disposable #3 blade and a stylet for placement of the endotracheal tube. This group is considered the "control group".
2. Intubation using the King Vision video-laryngoscope with the disposable #3 blade and the fiber-optic bronchoscope (aScope III). This group is considered the "interventional group".

When randomized to the "control group" (King Vision video-laryngoscope with #3 disposable blade and a stylet) the procedure sequence is as follows:

1. Standard anesthesia monitoring which includes but is not limited to ECG, pulse oximetry, capnography, blood pressure and temperature monitoring. Their head will be on an anesthesia pillow. This is all standard procedure.
2. Anesthesiologist will induced with Fentanyl (1-2 ug/kg), propofol (2-4 mg/kg). This is standard dosing.
3. Subjects will receive muscle relaxation using Rocuronium (0.6mg/kg) This is standard dosing.
4. The patient will be pre-oxygenated for 2-3 minutes with 100% oxygen by mask to achieve optimal oxygen saturation
5. One anesthesiologist will perform the intubation procedure using the King Vision video-laryngoscope with a #3 disposable blade and use a stylet to pre-form the endotracheal tube (ETT).
6. If the anesthesiologist's first attempt to intubate should fail the next attempt will use the standard Storz video-laryngoscope and a #4 reusable blade, a stylet to pre-form the endotracheal tube (ETT) and with external laryngeal pressure. (BURP: back, up, and rightward pressure)
7. The anesthesiologist may make a total of three attempts to intubate using the control group procedures. Each attempt should be less than 60 seconds and will be aborted if oxygen saturation falls below 90%. The patient will be pre-oxygenated by mask between each attempt.
8. After three failed attempts to intubate the anesthesiologist will use the interventional group method. Two anesthesiologists will be required to perform the intubation using the King Vision video-laryngoscope with a #3 disposable blade and the video bronchoscope (aScope III). The stylet will not be needed since the bronchoscope will be used to guide the endotracheal tube (ETT).
9. The video-laryngoscope will be used to visualize the glottis; the bronchoscope (aScope III) will be inserted underneath the epiglottis and advance to the carina under direct visualization. The endotracheal tube (ETT) will be threaded over the bronchoscope (aScope III) using the bronchoscope as a guide through the trachea.
10. Should the first attempt using the interventional method fail the next attempt will use the standard Storz video-laryngoscope and #4 reusable blade along with the video bronchoscope (aScope III)
11. There may be three attempts using the interventional method. Each attempt should be less than 60 seconds. If the oxygen saturation decreases below 90% the attempt should be aborted. The patient will be pre-oxygenated by mask between each attempt.
12. After three unsuccessful attempts the patient will be awaken and an "awake" intubation procedure will take place.
13. The anesthesiologist will note any bleeding occurring during the procedure. Bleeding will be assessed as minimal, moderate, and significant.
14. Study ends once the patient is intubated and breath sounds confirmed or when it is decided an "awake" intubation is needed.

When randomized to the "interventional" group. (King Vision video-laryngoscope and #3 disposable blade and the video-bronchoscope (aScope III) The sequence of procedures will be:

1. Standard anesthesia monitoring which includes but is not limited to ECG, pulse oximetry, capnography, blood pressure and temperature monitoring. Their head will be on an anesthesia pillow. This is all standard procedure.
2. Anesthesiologist will induced with Fentanyl (1-2 ug/kg), propofol (2-4 mg/kg). This is standard dosing.
3. Subjects will receive muscle relaxation using Rocuronium (0.6mg/kg)This is standard dosing.
4. The patient will be pre-oxygenated for 2-3 minutes with 100% oxygen by mask to achieve optimal oxygen saturation
5. Two anesthesiologist will perform the procedure
6. The video-laryngoscope will be used to visualize the glottis; the bronchoscope (aScope III) will be inserted underneath the epiglottis and advance to the carina under direct visualization. The endotracheal tube (ETT) will be threaded over the bronchoscope (aScope III) using the bronchoscope as a guide through the trachea.
7. Should the first attempt fail to intubate the patient the next attempt will use the Storz video- laryngoscope with a #4 reusable blade with the video-bronchoscope (aScope III)
8. A total of three attempts may be made using the interventional method. Each attempt should be less than 60 seconds and aborted if the oxygen saturation falls below 90%. The patient will be pre-oxygenated by mask with 100% oxygen between each attempt.
9. If failure to intubate should occur the patient will be awaken and an "awake" intubation will be performed.
10. The anesthesiologist will note any bleeding occurring during the procedure. Bleeding will be assessed as minimal, moderate, and significant.
11. The study will end with successful intubation and confirmation of breath sounds or when it is determined an "awake" intubation is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patient will be eligible for the trial if they:

  1. Have a tumor of the oral cavity, pharynx or larynx and are scheduled for biopsy or resection requiring intubation of the trachea
  2. Are 18 years or older
  3. Sign the approved inform consent

Exclusion Criteria:

* Patients will be excluded from the study if:

  1. Cannot lie down flat without suffering dyspnoea
  2. Stridor
  3. Full stomach
  4. Hiatal hernia
  5. Severe Gastroesophageal Reflux Disease (GERD) defined as already on a protein pump inhibitor and continues to have daily regurgitation
  6. Require rapid sequence intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Time to successful intubation | From time full relaxation is achieved to time the patients is successfully intubated confirmed by breath sounds over a period of up to ten minutes
  measured in seconds

SECONDARY OUTCOMES:
Conversion from control group to intervention group | From the time full relaxation is achieved until the subject is successfully intubated confirmed by breath sounds over a period of up to ten minutes
  Number of subjects randomized to control group who require to be treated with the method of the intervention group
Number of intubation attempts until successful | From the time full relaxation is achieved until the time the subject is intubated; confirmed with breath sounds over a period of up to ten minutes
  whole numbers of attempts

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Lenhardt, MD MBA, Principal Investigator — University of Louisville 530 South Jackson Street Louisville, KY 40202
Locations (1):
- University of Louisville Medical School, Department of Anesthesiology and Perioperative Medicine, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided
individual patients data will not be shared. Results or the studies findings will be published

REFERENCES:
- [Background] Juneja R, Lacey O. Anaesthesia for head and neck cancer surgery. Curr Anaesth Crit Care 2009;20:28-32.
- [Background] Stacey M, Rassam S, Sivasankar R, Hall J. Difficulty in advancing a tracheal tube over a fibreoptic bronchoscope: more solutions. Br J Anaesth. 2005 Jul;95(1):112. doi: 10.1093/bja/aei570. No abstract available. PMID 15941739
- [Background] Cooper RM. Use of a new videolaryngoscope (GlideScope) in the management of a difficult airway. Can J Anaesth. 2003 Jun-Jul;50(6):611-3. doi: 10.1007/BF03018651. PMID 12826557
- [Background] Doyle DJ. GlideScope-assisted fiberoptic intubation: a new airway teaching method. Anesthesiology. 2004 Nov;101(5):1252. doi: 10.1097/00000542-200411000-00046. No abstract available. PMID 15505482
- [Background] Turkstra TP, Harle CC, Armstrong KP, Armstrong PM, Cherry RA, Hoogstra J, Jones PM. The GlideScope-specific rigid stylet and standard malleable stylet are equally effective for GlideScope use. Can J Anaesth. 2007 Nov;54(11):891-6. doi: 10.1007/BF03026792. PMID 17975233
- [Background] Turkstra TP, Jones PM, Ower KM, Gros ML. The Flex-It stylet is less effective than a malleable stylet for orotracheal intubation using the GlideScope. Anesth Analg. 2009 Dec;109(6):1856-9. doi: 10.1213/ANE.0b013e3181bc116a. PMID 19923515
- [Background] Knill RL. Difficult laryngoscopy made easy with a "BURP". Can J Anaesth. 1993 Mar;40(3):279-82. doi: 10.1007/BF03037041. PMID 8467551
- [Background] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827
- [Background] Janda M, Scheeren TW, Noldge-Schomburg GF. Management of pulmonary aspiration. Best Pract Res Clin Anaesthesiol. 2006 Sep;20(3):409-27. doi: 10.1016/j.bpa.2006.02.006. PMID 17080693
- [Background] Fasting S, Gisvold SE. Serious intraoperative problems--a five-year review of 83,844 anesthetics. Can J Anaesth. 2002 Jun-Jul;49(6):545-53. doi: 10.1007/BF03017379. PMID 12067864
- [Result] Siu LW, Mathieson E, Naik VN, Chandra D, Joo HS. Patient- and operator-related factors associated with successful Glidescope intubations: a prospective observational study in 742 patients. Anaesth Intensive Care. 2010 Jan;38(1):70-5. doi: 10.1177/0310057X1003800113. PMID 20191780
- [Result] Van Zundert AA, Hermans B, Kuczkowski KM. Successful use of a videolaryngoscope in a patient with carcinoma of the oropharynx and obstructed airway. Minerva Anestesiol. 2009 Jul-Aug;75(7-8):475-6. No abstract available. PMID 19571781
- [Result] Lenhardt R, Burkhart MT, Brock GN, Kanchi-Kandadai S, Sharma R, Akca O. Is video laryngoscope-assisted flexible tracheoscope intubation feasible for patients with predicted difficult airway? A prospective, randomized clinical trial. Anesth Analg. 2014 Jun;118(6):1259-65. doi: 10.1213/ANE.0000000000000220. PMID 24842175